CLINICAL TRIAL: NCT05953584
Title: A Phase 2 Open-label Study to Evaluate the Activity of Etavopivat on Transcranial Doppler Velocities in Pediatric Patients With Sickle Cell Disease Who Are at Increased Risk for Primary Stroke
Acronym: HIBISCUS 3
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Forma Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Organization: Novo Nordisk A/S (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4202-HEM-204; PACTR202301655446404 (Registry Identifier: Pan African Clinical Trial Registry)
Record Dates: First submitted 2023-07-11; First posted 2023-07-20 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Hydroxyurea

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Etavopivat (Experimental): Participants will receive Etavopivat 400 mg once daily (QD) orally.
  Interventions: Drug: Etavopivat
- Etavopivat with HU (Experimental): Participants will receive Etavopivat 400 mg QD orally in combination with HU. The dose of HU (mg/kg) will be stable (no more than a 20% change in dosing except for weight-based changes) during the study, in the opinion of the Investigator.
  Interventions: Drug: Etavopivat; Drug: Hydroxyurea

INTERVENTIONS:
Drug: Etavopivat — Participants will receive a dose of 400 mg (two 200 mg oral tablets) etavopivat once daily.
Drug: Hydroxyurea — Participants will receive a stable dose of HU.
  Arms: Etavopivat with HU

SUMMARY:
The study will test a new medicine, etavopivat, for sickle cell disease and see if it is safe and help-ful for participants with sickle cell disease who are at an increased risk of stroke. Participants will be divided into two cohorts depending on their transcranial doppler (TCD) ultrasound results and whether or not they receive hydroxyurea (medication that they may already be taking). In one cohort, participants with conditional transcranial doppler (TCD) or participants with abnormal TCD who are not able to receive hydroxyurea will be included. The study doctor will determine if the TCD result is conditional or abnormal. In another cohort, participants with conditional TCD or participants with abnormal TCD who are receiving a stable dose of hydroxyurea will be included. The study doctor will determine if the TCD result is conditional or abnormal. The participant will start a 52-week (1 year) treatment period. The participant will take 400 milligrams (mg) of etavopivat once a day for the 52 weeks. The dose of 400 mg will be taken as 2 tablets by mouth, each containing 200 mg of etavopivat. Etavopivat may be taken with or without food. Each dose should be taken with a glass of water. As part of the study, the participants will be asked to visit the clinic frequently. The participant will have the opportunity to participate in a 48-week optional extension treatment period. The optional extension treatment period will allow continued as-sessment of safety of etavopivat in paediatric patients. At the end of the study, if deemed appro-priate the participant, the caregiver, and the study doctor, the participant may be offered the op-portunity to participate in a separate study to continue receiving etavopivat. If/when this separate study becomes available, the participant may only transfer to the new study after completion of the 52-week primary treatment period and at any time during the 48-week optional extension treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Patient's parent, legal guardian, or legal representative has provided documented informed consent and patients have provided age-appropriate assent

   Age:
2. 12 to 16 years of age (inclusive) at time of screening

   Type of Participant and Disease Characteristics:
3. Confirmed diagnosis of SCD

   • Documentation of any SCD genotype (e.g. HbSS, HbSβ0 -thalassemia) based on prior history of laboratory testing. Molecular genotyping is not required. SCD genotype may be determined from the results of Hb electrophoresis, high-performance liquid chromatography, or similar testing.
4. TAMMV greater than or equal to (≥) 170 cm/s in the ICA and/or MCA during the Screening Period and confirmed on 2 occasions and without history of primary ischemic or hemorrhagic stroke, transient ischemic attack, or severe central nervous system (CNS) vasculopathy on magnetic resonance angiography (MRA). This includes patients with cTCD (170-199 centimeter per second [cm/s]) or aTCD (≥ 200 cm/s). Patients with aTCD cohort must have refused transfusion therapy.
5. Hb ≥ 6 grams per deciliter (g/dL) and lesser than or equal to (≤) 9 g/dL at screening
6. For participants with aTCD and cTCD and already taking HU, the dose of HU milligram per kilogram (mg/kg) must be stable (no more than a 20% change in dosing except for weight-based changes) for at least 90 days prior to start of study treatment with no anticipated need for dose adjustments except for weight-based changes during the study, in the opinion of the Investigator.

   Sex and Contraceptive Requirements
7. Patients, who if female and of childbearing potential, are using acceptable methods of contraception and agree not to donate ova from study start to 90 days after the last dose of study drug, and who if male, are willing to use acceptable methods of contraception and agree not to donate sperm, from study start to 90 days after the last dose of study drug

Exclusion Criteria:

Medical Conditions

1. Female who is breast feeding or pregnant
2. History of seizure disorder
3. Prior overt stroke (a focal neurological deficit of acute onset) by history or significant concerns for history of overt stroke based on Screening MRL, history of transient ischemic attack, focal neurological deficit on standardized neurological examination, or concern for moderate or severe neurological deficit (which could be due to stroke) based on a positive "10 questions" screening. Patients with significant or suggestive severe CNS vasculopathy (ie, moya moya) of Grade 4 or higher based on MRA read locally.
4. Significant cytopenias (absolute neutrophil count [ANC] < 1.5 × 10^3/microliter (µL), platelets < 150,000/µL, reticulocytes < 80,000/µL)
5. Severe renal dysfunction (estimated glomerular filtration rate at the Screening visit; calculated by the local laboratory < 30 mL/min/1.73 m^2) or on chronic dialysis
6. Hepatic dysfunction characterized by alanine aminotransferase (ALT) > 4 × upper limit of normal (ULN) and/or direct bilirubin > 3 × ULN
7. Patients with clinically significant bacterial, fungal, parasitic, or viral infection requiring systemic therapy or history of such infections leading to significant neurological impairment:

   * Patients with acute bacterial, fungal, parasitic, or viral infection requiring systemic therapy should delay screening/enrollment until active therapy has been completed.
   * Patients with acute viral infections (eg, coronavirus disease 2019 [COVID-19]) should delay screening/enrollment until the acute infection has resolved.
   * Patients enrolled in areas where malaria is prevalent must be on malaria prophylaxis based on regional guidance and resistance results. Note: Infection prophylaxis is allowed (see concomitant medication restrictions).
8. Known human immunodeficiency virus (HIV) positivity
9. Known infection with hepatitis B virus (hepatitis B surface antigen [HepBsAg] and hepatitis B core antibody [HepBcAb] positive.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Estimated)
Dates: Start 2023-06-20 (Actual); Primary Completion 2027-09-20 (Estimated); Study Completion 2027-09-20 (Estimated)

PRIMARY OUTCOMES:
Change in the highest TAMMV in any of the L/R internal carotid artery [ICA] and L/R middle cerebral artery [MCA], whichever is highest, as measured by TCD | Baseline and Week 12

SECONDARY OUTCOMES:
Change in the highest TAMMV in any of the L/R internal carotid artery [ICA] and L/R middle cerebral artery [MCA], whichever is highest, as measured by TCD | Baseline, Weeks 2,4, 24 and 52
Incidence of conversion to normal (< 170 cm/s), conditionally abnormal (170-199 cm/s), and abnormal (≥ 200 cm/s) TCD velocities | Weeks 2, 4, 12, 24, and 52

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (9):
- India (5):
  - All India Institute of Medical Sciences (AIIMS), Raipur, Raipur, Chhattisgarh
  - All India Institute of Medical Sciences-Delhi, Delhi
  - Nirmal Hospital Pvt. Ltd., Gujarat
  - Suretech Hospital and Research Centre Ltd., Maharashtra
  - Indira Gandhi Government Medical College & Hospital, Nagpur
- Nigeria (3):
  - University of Ibadan, University College Hospital, Ibadan
  - Lagos University Teaching Hospital, Lagos, Lagos
  - Aminu Kano Teaching Hospital (AKTH), Tarauni
- Sultan Qaboos University Hospital, Muscat, Sultanet of Oman/Muscat/Al Khoud, Oman

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com